CLINICAL TRIAL: NCT04855695
Title: A Phase 1/2 Study of Acalabrutinib, Venetoclax, and Obinutuzumab in Patients With Relapsed/Refractory and Previously Untreated Mantle Cell Lymphoma
Brief Title: Avo In R/R And Previously Untreated MCL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Austin I Kim (Other)
Collaborators: Roche-Genentech (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Austin I Kim, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-040
Record Dates: First submitted 2021-04-11; First posted 2021-04-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Mantle Cell Lymphoma; Refractory Lymphoma
Keywords: Mantle Cell Lymphoma; Refractory Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma | interventions — acalabrutinib; venetoclax; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Acalabrutinib, Venetoclax, and Obinutuzumab (Experimental): The study will consist of 4 parts (Parts A, B, C, and D). In the relapsed/refractory (R/R) MCL setting (Part A), the phase 1 portion consists of a dose finding stage to determine the recommended phase 2 dose (RP2D). It will follow a 3+3 dose finding schema with a minimum of 6 participants. 11 participants will be enrolled in the Part A expansion cohort.
  Part B will enroll 24 participants with untreated mantle cell lymphoma who are transplant ineligible and/or TP53 mutated.
  Part C will enroll 12 participants with untreated mantle cell lymphoma who are transplant eligible and TP53 wild type.
  Part D will enroll 16 participants with untreated mantle cell lymphoma with a TP53 mutation determined by next generation sequencing, regardless of transplant eligibility.
  Each study drug is given according to a different schedule. Each treatment cycle lasts 28 days (4 weeks).
  * Acalabrutinib:
  * Obinutuzumab:
  * Venetoclax:
  Interventions: Drug: Acalabrutinib; Drug: Venetoclax; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Acalabrutinib — Each study drug is given according to a different schedule:
  Acalabrutinib: Oral, dosage per protocol, start cycle 1 and beyond according to schedule outlined in protocol
  Other Names: Calquence, Acalabrutinib maleate
Drug: Venetoclax — Venetoclax: oral. daily, dosage per protocol, start cycle 3 and beyond according to schedule outlined in protocol
  Other Names: Venclexta
Drug: Obinutuzumab — Obinutuzumab: intravenous infusion, dosage per protocol, drug during cycles 2 and beyond according to schedule outlined in protocol
  Other Names: Gazyva

SUMMARY:
This research study is evaluating the combination of three drugs - acalabrutinib, venetoclax, and obinutuzumab - as a possible treatment for relapsed or refractory and untreated mantle cell lymphoma (MCL).

The names of the study drugs involved in this study are:

* Acalabrutinib
* Venetoclax
* Obinutuzumab

DETAILED DESCRIPTION:
This is an open-label, investigator-initiated, single-arm, multi-cohort phase 1/2 study to assess the safety and efficacy of the combination of acalabrutinib, venetoclax, and obinutuzumab (AVO) in relapsed/refractory (R/R) and untreated mantle cell lymphoma (MCL).

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

The names of the study drugs involved in this study are:

* Acalabrutinib
* Venetoclax
* Obinutuzumab

Participants will receive study treatment for as long as there are no serious side effects and the disease does not get worse. Participants will be followed for 5 years.

It is expected that 72 people will take part in this research study.

This is a Phase I/II clinical trial. Phase I clinical trials test the safety of investigational drugs and also tries to define the appropriate dose of investigational drugs to use for further studies. "Investigational" means that the drugs are being studied.

* The U.S. Food and Drug Administration (FDA) has not approved venetoclax and obinutuzumab for this specific disease but it has been approved for other uses.
* The U.S. Food and Drug Administration (FDA) has approved acalabrutinib as a treatment option for this disease.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study:
* Participants must have histologically determined mantle cell lymphoma with pathologic review at the participating institutions, that has either:

  * Relapsed or primary refractory after at least one line of therapy including anti-CD20 monoclonal antibody treatment (part A) or; Had no previous anti-lymphoma therapy other than corticosteroids or radiotherapy (parts B, C, and D).
  * Participants in part A, relapsed or refractory following prior therapy, may have had a prior autologous or allogeneic stem cell transplant and may have been treated with chimeric antigen receptor T-cells (CAR T-cells).
* Participants in parts B, C, and D, without prior anti-lymphoma therapy, must require treatment as defined by any of the following criteria:

  * Symptomatic adenopathy or splenomegaly
  * Local symptoms due to extranodal disease
  * Organ function impairment due to disease involvement, including cytopenias due to marrow involvement (WBC <1.5x109/L; absolute neutrophil count [ANC] <1.0x109/L, Hgb <10g/dL; platelets <100x109/L)
  * Presence of systemic B symptoms (fever, drenching night sweats, or unintentional weight loss ≥ 10% body weight over previous 6 months) or functionally significant fatigue
* Participants in part B without prior anti-lymphoma therapy should be deemed to be ineligible for autologous stem cell transplant by the treating physician and/or have a TP53 mutation detected by next generation sequencing at a variant (mutant) allele fraction above the validated threshold for calling a new variant or high TP53 expression on immunohistochemistry (>50% positive lymphoma cells)
* Participants in part C without prior anti-lymphoma therapy should be deemed to be eligible for autologous stem cell transplant by the treatment physician and have no evidence of TP53 mutation (TP53 wild type) detected by next generation sequencing and no evidence of high TP53 expression on immunohistochemisty
* Participants in part D without prior anti-lymphoma therapy must have a TP53 mutationdetected by next generation sequencing at a variant (mutant) allele fraction above thevalidated threshold for calling a new variant
* Participants in parts B, C, and D must have an archived formalin-fixed paraffin-embedded (FFPE) tumor tissue specimen from the original diagnostic biopsy and peripheral blood available for submission to Adaptive Biotechnologies for ClonoSEQ®ID molecular marker identification of a unique clonal immunoglobulin DNA sequence. Only those participants in parts B and C who have a molecular marker identified from the peripheral blood will be eligible for minimal residual disease (MRD) driven treatment interruptions.
* Participants in parts B, C, and D who do not have a molecular marker identified by ClonoSEQ from the peripheral blood will be deemed to be MRD indeterminate and are not eligible for peripheral blood MRD driven treatment interruptions. These participants will be able to enroll in the study assuming all other eligibility criteria are met but will receive 7 cycles of AVO combination therapy followed by 17 cycles of acalabrutinib and venetoclax therapy (24 total cycles of AV) and 2 years of maintenance obinutuzumab for a total of 31 cycles of therapy.
* Measurable disease with a lymph node or tumor mass ≥ 1.5 cm in at least one dimension by CT, PET/CT, or MRI. Patients without measurable disease will be eligible if they have marrow involvement and cytopenias related to their lymphoma (hemoglobin <10 g/dL, absolute neutrophil count < 1.0 x 109/L, or platelets < 100 x 109/L) OR symptomatic splenomegaly > 15cm in craniocaudal diameter.
* Age ≥ 18 years.
* ECOG performance status ≤2 (Karnofsky ≥60%)
* Participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 750 cells/mm3 (0.75 x109/L) unless due to marrow involvement by lymphoma in which case ANC must be ≥ 500 cells/mm3 (0.5x109/L)
  * Platelet count without transfusional support must be ≥ 75,000 cells/mm3 (75 x109/L), unless due to marrow involvement by lymphoma, in which case platelets must be ≥ 50,000 cells/mm3 (50 x109/L)
  * Hemoglobin without transfusional support must be ≥ 8.0 g/dL (80 g/L) unless due to marrow involvement by lymphoma, in which case hemoglobin must be ≥ 7.0 g/dL (70 g/L)
  * Creatinine clearance (CrCl) ≥ 50 ml/min using 24-hour urine collection for creatinine clearance or calculated CrCl or calculated glomerular filtration rate (GFR) ≥ 50 ml/min/1.73 m2 using the CKD-EPI equation
  * Total bilirubin ≤ 2 times the upper limit of normal, unless there is disease involvement of the liver, hemolysis, or a known history of Gilbert's disease, in which case direct bilirubin must be ≤ 3 times the upper limit of normal
  * AST and ALT ≤ 2.5 times the upper limit of normal, unless documented liver involvement by lymphoma, in which case AST and ALT must be ≤ 5 times the upper limit of normal
  * PT/INR ≤ 2 times the upper limit of normal and PTT ≤ 2 times the upper limit of normal
* Willingness to provide pre-treatment bone marrow (or recent archival w/o intervening therapy) and on-treatment bone marrow and peripheral blood samples
* The effects of the study drugs on the developing human fetus are unknown. Women of child-bearing potential must agree to remain abstinent or use highly effective contraception (defined as contraceptive measures that result in a failure rate of <1% per year) during the treatment period and for at least 2 days after the last dose of acalabrutinib, 90 days after the last dose of venetoclax or 18 months after the last dose of obinutuzumab, whichever is longer. Men with female sexual partners of childbearing potential should agree to remain abstinent or use contraceptive measures which include a condom plus an additional contraceptive method that together result in a failure rate of <1% per year during the treatment period and for at least 90 days after the last dose of venetoclax or 6 months after the last dose of obinutuzumab, whichever is longer. Men should refrain from donating sperm during the same period. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not eligible for admission into the study:
* Participants who have progressed or relapsed after receiving either a BTK inhibitor or BCL2 inhibitor.
* Participants who are receiving any other investigational agents, or have received investigational agents within 4 weeks (or 3 half-lives, whichever is longer) of beginning treatment.
* Concurrent systemic immunosuppressant therapy (e.g., cyclosporine A, tacrolimus, etc., within 28 days of the first dose of study drug or chronic administration of >20 mg/day of prednisone equivalent corticosteroid within 7 days of the first dose)

  -- Note: Glucocorticoids for lymphoma symptom palliation are allowed but must be discontinued at time of initiation of protocol therapy.
* History of severe allergic reactions attributed to compounds of similar chemical or biologic composition to obinutuzumab, venetoclax, or acalabrutinib. Patients with reactions to other CD20 monoclonal antibodies (e.g. rituximab, ofatumumab) are not excluded if they were able to eventually tolerate treatment in an outpatient setting without grade 2 or higher infusion reactions.
* Participants who have a history of other malignancies except:

  * Malignancy treated with curative intent and with no known active disease present and felt to be at low risk for recurrence by treating physician. Current adjuvant hormonal therapy for disease treated with curative intent is permissible.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated carcinoma in situ without evidence of disease.
  * Low-risk prostate cancer on active surveillance
  * Other exceptions may be made after consultation with the study chair
* Participants with known leptomeningeal or brain metastases. Imaging or spinal fluid analysis to exclude CNS involvement is not required, unless there is clinical suspicion by the treating investigator.
* Participants who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, participants who have not adequately recovered from the side effects of any major surgery (defined as requiring general anesthesia), or participants that may require major surgery during the course of the study.
* Vaccinated with live, attenuated vaccines within 28 days of study entry or need for live virus vaccines at any time during study period.
* Patients with human immunodeficiency virus (HIV) or active hepatitis C virus (HCV) or hepatitis B virus (HBV) infection. HIV-positive participants are ineligible because of the potential for pharmacokinetic interactions between certain components of anti-retroviral therapy and venetoclax. Patients who are positive for hepatitis B core antibody or hepatitis B surface antigen must have a negative polymerase chain reaction (PCR) result before enrollment. Those who are PCR positive will be excluded. Those who are positive for either hepatitis B surface antigen and/or hepatitis B core antibody but negative for HBV DNA will be managed. Patients who are positive for HCV antibody must be negative for HCV by polymerase chain reaction (PCR) to be eligible for study participation.
* Ongoing or recent infection requiring intravenous antimicrobials at time of screening. Patients with ongoing use of prophylactic antibiotics are eligible as long as there is no evidence of active infection and the antibiotic is not included on the list of prohibited medications.
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements, compromise the subject's safety, or put the study outcomes at undue risk.
* Lactating or pregnant women are excluded from this study because venetoclax has been shown to decrease implantation, litter size, live fetuses, and fetal body weight in animal models. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with venetoclax, breastfeeding should be discontinued if the mother is treated with venetoclax. These potential risks may also apply to other agents used in this study.
* Known bleeding disorders (e.g. von Willebrand's disease) or hemophilia.
* Presence of a bleeding gastrointestinal ulcer diagnosed by endoscopy within 3 months prior to enrollment.
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
* Participants who require warfarin or other vitamin K antagonists for anticoagulation (other anticoagulants are allowed).
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization. Patients with atrial fibrillation are allowed as long as they are adequately rate controlled.
* Participants who require concurrent treatment with strong CYP3A inhibitors or strong CYP3A inducers are excluded from the study. If patients are receiving strong CYP3A inhibitors/inducers at time of screening but do not require continuous administration of these agents, these patients are eligible if there is a 7-day washout period between discontinuation of the strong CYP3A inhibitor/inducer and initiation of the first study drug, acalabrutinib.
* Participants who require concurrent treatment with P-gp inhibitors or narrow therapeutic index P-gp substrates are excluded from the study. If patients are receiving P-gp inhibitors or narrow therapeutic index P-gp substrates at time of screening but do not require continuous administration of these agents, these patients are eligible if there is a 7-day washout period between discontinuation of the P-gp inhibitor and initiation of venetoclax.
* Unable to swallow capsules, a large number of tablets, or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel if thought by the investigator to compromise systemic absorption, active, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.
* Significant co-morbid condition or disease which in the judgment of the Principal Investigator would place the participant at undue risk or interfere with the study.
* History of or ongoing confirmed progressive multifocal leukoencephalopathy (PML).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose for acalabrutinib | 5 months
  The RP2D will be defined as the highest dose level for which there are no more than 1/6 DLTs observed.
Complete Remission Rate | 7 Months
  Complete remission (CR) rate after 7 cycles of treatment with AVO in treatment naïve (TN) transplant ineligible MCL and TN transplant-eligible, TP53 mutated MCL, cohort B. CR rate after 7 cycles of treatment with AVO in TN TP53-mutated MCL, expansion cohort D.
  Complete remission (CR) is defined radiographically using 2014 Lugano criteria and a negative bone marrow biopsy by histology, immunohistochemistry, and flow cytometry, if bone marrow was initially involved by MCL at screening. CR, a primary endpoint measured after 7 cycles of AVO, does not incorporate minimal residual disease (MRD) testing
MRD negative complete remission rate | 7 months
  Minimal residual disease (MRD) negative (<1 in 106 cells) CR rate after 7 cycles of treatment with AVO in TN transplant-eligible, TP53 wild type MCL, cohort C

SECONDARY OUTCOMES:
CR rate after 7 cycles of treatment with AVO in participants with TN TP53-mutated MCL in cohort B and expansion cohort D | 7 cycles
  Complete remission (CR) is defined radiographically using 2014 Lugano criteria and a negative bone marrow biopsy by histology, immunohistochemistry, and flow cytometry, if bone marrow was initially involved by MCL at screening. CR, a primary endpoint measured after 7 cycles of AVO, does not incorporate minimal residual disease (MRD) testing
Complete Remission (CR) rate after 7 cycles in the entire study population | 7 months
  Complete remission (CR) is defined radiographically using 2014 Lugano criteria and a negative bone marrow biopsy by histology, immunohistochemistry, and flow cytometry, if bone marrow was initially involved by MCL at screening. CR, a primary endpoint measured after 7 cycles of AVO, does not incorporate minimal residual disease (MRD) testing
CR rate after 7 cycles cohort A and C | 7 Months
  Complete remission (CR) is defined radiographically using 2014 Lugano criteria and a negative bone marrow biopsy by histology, immunohistochemistry, and flow cytometry, if bone marrow was initially involved by MCL at screening. CR, a primary endpoint measured after 7 cycles of AVO, does not incorporate minimal residual disease (MRD) testing
Partial Response (PR) Rate after 7 cycles | 7 months
  2014 Lugano Criteria
Stable Disease Rate after 7 cycles | 7 months
  Stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started, including the baseline measurements.
Progressive Disease Rate after 7 Cycles | 7 months
  Lugano 2014 criteria
Progression Free Survival-Median | Up to 5 Years
  Kaplan Meier Progression-Free Survival (PFS) is defined as the time from randomization (or registration) to the earlier of progression or death due to any cause.
  Participants alive without disease progression are censored at date of last disease evaluation
Progression Free Survival | Up to 5 years
  Kaplan Meier Progression-Free Survival (PFS) is defined as the time from randomization (or registration) to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation
Overall Survival | Up to 5 years
  Kaplan Meier- Overall Survival (OS) is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive.
Overall Survival-Median | Up to 5 years
  Kaplan Meier Overall Survival (OS) is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive.
Rate of peripheral blood MRD-negativity after 7 cycles | 7 months
  Minimal residual disease (MRD) negativity is defined as 0 residual clonal cells per 1 x 106 nucleated cells in the peripheral blood assessed by the clonoSEQ® assay. The clonoSEQ assay uses next generation sequencing (NGS) to identify rearranged IgH (VDJ), IgH (DJ), IgK, and IgL receptor gene sequences, as well as translocated BCL1/IgH (J) sequences in a sample
Time to Minimal Residual Disease (MRD)-positive disease recurrence in the peripheral blood | Up to 8 months
  Time to MRD-positive disease recurrence, in patients who have achieved MRD negativity
Time to clinical disease progression | Up to 5 years
  Time to Progression (TTP) is defined as the time from randomization (or registration) to progression, or censored at date of last disease evaluation for those without progression reported
Rate of infusion related reactions | Up to 5 years
  Some participants may develop hypersensitivity or other infusion-related reactions (IRRs) to obinutuzumab, pre-medication is recommended to reduce the risk of infusion reactions. Premedication will be given as outlined in protocol. Cycle numbers are specific to this trial
Rate of tumor lysis syndrome | 7 Months
  criteria of laboratory TLS or clinical TLS according to the Cairo-Bishop definition of TLS
Rate of therapy discontinuation | 10 Months
  descriptive analysis of rates of therapy discontinuation after 10 cycles will be performed, with subjects grouped by reasons for discontinuation (e.g. achievement of MRD-negative CR, progressive disease, or intolerability). Rates of discontinuation of individual components of the regimen will also be included in this analysis.
Number of Participants with Treatment Related Adverse Events CTCAE 5.0 criteria | up to 30 days after the last dose of study treatment or until resolution of toxicity to grade 1 or baseline, whichever occurs last up to 5 years
  Grade 3 and higher toxicities, both regardless of attribution, and at least possibly attributed to the study treatment
  * Grade 2 or higher toxicity at least probably related to study treatment
  * Adverse events leading to discontinuation due to toxicity
  NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Austin I Kim, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - University of Chicago Medical Center, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu